CLINICAL TRIAL: NCT00494520
Title: Learning Paradigms in Aphasia Rehabilitation
Brief Title: Cognitive Therapy to Improve Word Finding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DC006934-01 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2014-04

CONDITIONS: Anomia; Aphasia; Traumatic Brain Injury; Cerebrovascular Accident
Keywords: Anomia; Aphasia; Traumatic Brain Injury; Cerebrovascular Accident
MeSH Terms: conditions — Anomia; Aphasia; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Errorful training condition (Experimental): A type of anomia rehabilitation paradigm which allows for errors. The intervention involves providing minimal auditory cues to allow for errors in picture naming.
  Interventions: Procedure: Errorful training condition
- Errorless training condition (Experimental): A type of anomia rehabilitation paradigm in which the situation surrounding the performance of the desired task (i.e., picture naming) is controlled to prevent errors. The intervention involves providing maximal auditory cues to prevent errors in picture naming.
  Interventions: Procedure: Errorless training condition

INTERVENTIONS:
Procedure: Errorful training condition — Errorful training condition: Participant saw a picture and named it without any cues. If an error was produced, the cue with the least amount of information was provided (e.g. for "pumpkin", "pu"). Cues with increasing information were provided until the picture was correctly named (e.g. for "pumpkin": "pump", "pumpki", then "pumpkin"). Once the correct name was provided, the trial ended.
  Arms: Errorful training condition
Procedure: Errorless training condition — Errorless learning (EL) condition: Participant saw a picture with its name, and repeated the word. The participant continued to name the picture as the auditory cues provided less and less of the word (e.g. for "banana" she would hear "banan", "bana" then "ba" and finally no cue). If an error was produced at any stage, the whole word was presented, the participant repeated it, and the trial ended.
  Arms: Errorless training condition

SUMMARY:
Adults who sustain brain damage due to stroke, traumatic injury or surgery may develop difficulty finding words. This study compares the effectiveness of two behavior-based programs to improve picture naming ability in these individuals.

DETAILED DESCRIPTION:
Difficulty finding words is common in patients with aphasia subsequent to left hemisphere stroke. This study will compare two cognitive therapies for the treatment of acquired word finding difficulties. The therapies use different types of cues. All participants will receive both therapies. Participants in this study will undergo a comprehensive and detailed assessment of language and other cognitive skills. The two treatments will be compared for their efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Word finding difficulty subsequent to stroke, traumatic brain injury, brain surgery or other brain damage occuring at least 6 month prior to participation
* Ability to attend 2 sessions per week for several months at Georgetown University in Washington, DC

Exclusion Criteria:

* History of learning disabilities
* Best corrected vision less than 20/40
* Corrected hearing within functional limits
* Less than 10 years formal education
* Significant memory or comprehension problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2004-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improved picture naming of trained words. | Following conclusion of word treatment.
  Overall accuracy of named trained items

SECONDARY OUTCOMES:
Improved picture naming of trained words. | At 6 months after conclusion of word treatment
  Overall accuracy of named trained items
Improved picture naming of untrained words. | Following conclusion of word treatment.
  Overall accuracy of named untrained items
Improved picture naming of untrained words. | At 6 months after conclusion of word treatment
  Overall accuracy of named untrained items

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda B. Friedman, Ph.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cognitive Neuropsychology Lab at Georgetown University Medical Center — http://www9.georgetown.edu/faculty/friedmar/index.html